CLINICAL TRIAL: NCT04583995
Title: A Phase 3, Randomised, Observer-Blinded, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of a SARS-CoV-2 Recombinant Spike Protein Nanoparticle Vaccine (SARS-CoV-2 rS) With Matrix-M1™ Adjuvant in Adult Participants 18-84 Years of Age in the United Kingdom
Brief Title: A Study Looking at the Effectiveness, Immune Response, and Safety of a COVID-19 Vaccine in Adults in the United Kingdom
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019nCoV-302
Record Dates: First submitted 2020-10-09; First posted 2020-10-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — NVX-CoV2373 adjuvated lipid nanoparticle; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: SARS-CoV-2 rS/Matrix-M1 Adjuvant (Experimental): 2 doses of 5 µg SARS-CoV-2 rS + 50 µg Matrix-M1 adjuvant (co-formulated), 1 dose each on Days 0 and 21.
  Interventions: Biological: SARS-CoV-2 rS/Matrix M1-Adjuvant
- Cohort 1: Placebo (Placebo Comparator): 2 doses of Placebo (Saline), 1 dose each on Days 0 and 21.
  Interventions: Other: Placebo
- Cohort 2: SARS-CoV-2 rS/Matrix-M1 Adjuvant Plus Licensed Seasonal Flu Vaccine (Experimental): 2 doses of 5 µg SARS-CoV-2 rS + 50 µg Matrix-M1 adjuvant (co-formulated), 1 dose each on Days 0 and 21. 1 dose of licensed seasonal flu vaccine on Day 0.
  Interventions: Biological: SARS-CoV-2 rS/Matrix M1-Adjuvant; Biological: Licensed seasonal influenza vaccine
- Cohort 2: Placebo Plus Licensed Seasonal Flu Vaccine (Placebo Comparator): 2 doses of Placebo (Saline), 1 dose each on Days 0 and 21. 1 dose of licensed seasonal flu vaccine on Day 0.
  Interventions: Other: Placebo; Biological: Licensed seasonal influenza vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 rS/Matrix M1-Adjuvant — Alternating intramuscular (deltoid) injections of SARS-CoV-2 rS co-formulated with Matrix-M1 adjuvant (0.5 mL) on Days 0 and 21.
  Other Names: NVX-CoV2373
  Arms: Cohort 1: SARS-CoV-2 rS/Matrix-M1 Adjuvant; Cohort 2: SARS-CoV-2 rS/Matrix-M1 Adjuvant Plus Licensed Seasonal Flu Vaccine
Other: Placebo — Alternating intramuscular (deltoid) injections of placebo (0.5 mL) on Days 0 and 21.
  Other Names: Sodium chloride 0.9% (BP, sterile)
  Arms: Cohort 1: Placebo; Cohort 2: Placebo Plus Licensed Seasonal Flu Vaccine
Biological: Licensed seasonal influenza vaccine — Single intramuscular injection of licensed seasonal flu vaccine, administered ideally in opposite deltoid to SARS-CoV-2 rS with Matrix-M1 adjuvant or placebo injection on Day 0.
  Arms: Cohort 2: Placebo Plus Licensed Seasonal Flu Vaccine; Cohort 2: SARS-CoV-2 rS/Matrix-M1 Adjuvant Plus Licensed Seasonal Flu Vaccine

SUMMARY:
This is a study to evaluate the efficacy, immune response, and safety of a coronavirus disease 2019 (COVID-19) vaccine called SARS-CoV-2 rS with Matrix-M1 adjuvant in adults aged 18-84 years in the United Kingdom. A vaccine causes the body to have an immune response that may help prevent the infection or reduce the severity of symptoms. An adjuvant is something that can make a vaccine work better. This study will look at the protective effect, body's immune response, and safety of SARS-CoV-2 rS with Matrix-M1 adjuvant in the study population. Participants in the study will randomly be assigned to receive SARS-CoV-2 rS with Matrix-M1 adjuvant or placebo. Each participant in the study will receive a total of 2 intramuscular injections over the course of the study. Approximately 15,000 participants will take part in the study. The first approximately 400 participants who meet additional criteria will receive a flu vaccine, in addition to the SARS-CoV-2 rS vaccine or placebo, as part of a sub-study.

An effort will be made to enroll a target of at least 25% of participants who are ≥ 65 years of age, as well as prioritizing other groups that are most affected by COVID-19, including racial and ethnic minorities.

Unblinding of treatment assignment may occur in order to allow a participant to make an informed decision regarding receipt of an already approved or deployed SARS-CoV-2 vaccine. Participants who choose to receive an approved or deployed SARS-CoV-2 vaccine as per UK government guidance will be encouraged to remain in the study for scheduled safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with all study requirements.
* Willing to allow investigators to discuss medical history with their General Practitioner and access all relevant medical records.
* Willing and able to give informed consent.
* Women of child-bearing potential must agree not to have sexual intercourse with men, or must consistently use an agreed method of contraception, from at least 28 days prior to enrolment in the study, through 3 months after the last vaccination.
* Room air oxygen saturation > 95% at Screening/Day 0.
* Seasonal Flu Vaccine Co-Administration Sub-Study only: Participant should not have received a current season flu vaccine, should have no reason why the specific sub-study flu vaccine cannot be administered, and should not have any prior history of allergy or severe reaction to seasonal flu vaccines.

Exclusion Criteria:

* Participation in other COVID-19 vaccine or preventative drug trials for the duration of the study.
* Future participation in any blood tests for the duration of the study where participants are informed of their levels of COVID-19 antibodies or antigens.
* Participation in any trial involving an investigational drug, biologic or device within 45 days prior to the first study vaccination.
* History of laboratory-confirmed COVID-19 infection any time prior to first study vaccination.
* Receipt of any immunoglobulins and/or any blood products within 3 months prior to planned administration of study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient state. Chronic administration (defined as more than 14 continuous days) of immunosuppressant medication within the past 3 months, except topical steroids or short-term oral steroids (course lasting ≤ 14 days). Note: An immunosuppressant dose of glucocorticoid is defined as a systemic dose ≥ 10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted if other chronic disease conditions do not exclude a participant from the study.
* History of allergic disease or reactions likely to be made worse by any component of the study vaccines.
* History of anaphylaxis to any prior vaccine.
* Pregnancy, breast-feeding or willingness/intention to become pregnant within 3 months following the last study vaccination.
* Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ.
* Bleeding disorder, or prior history of significant bleeding or bruising following intramuscular injections or venepuncture (e.g. to draw blood for tests).
* Continuous use of anticoagulants or anti-platelet agents. Note: The preventative use of ≤ 325 mg of aspirin per day is permitted.
* Suspected or known current alcohol or drug dependency.
* Study team member or first-degree relative of any study team member (inclusive of sponsor, contract research organization (CRO), and site personnel involved in the study).
* Participants having any current workup of undiagnosed illness within 8 weeks prior to start of study which could lead to new condition or diagnosis.
* Received any live vaccine within 4 weeks or any vaccine (excluding flu) within 2 weeks prior to first study vaccination; or any licensed flu vaccine within 1 week prior to first study vaccination or plans to receive any vaccine from these time periods until 28 days after the second study vaccination.
* Have clinically significant chronic cardiovascular, endocrine (hormones), gastrointestinal, hepatic (including hepatitis B and C), renal (kidney), neurological, respiratory, psychiatric or other medical disorders not excluded by other exclusion criteria, that are assessed by the investigator as being clinically unstable within the prior 4 weeks as evidenced by: a) Hospitalisation for the condition, including day surgical interventions; b) New significant organ function deterioration; or c) Needing addition of new treatments or major dose adjustments of current treatments (mild or moderate well-controlled comorbidities are allowed).
* History of chronic neurological disorders that have required prior specialist physician review for diagnosis and management (such as multiple sclerosis, dementia, transient ischemic attacks, Parkinson's disease, degenerative neurological conditions, and neuropathy) or a history of stroke or previous neurological disorder within 12 months with residual symptoms. Participants with a history of migraine or chronic headaches or nerve root compression that have been stable on treatment for the last 4 weeks are not excluded.
* Any autoimmune disease/condition (iatrogenic or congenital).
* Any other significant disease, disorder or finding that, in the opinion of the investigator, may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study, or impair interpretation of the study data.
* Participant requires the use of continuous oxygen therapy or any oxygen therapy while awake or is anticipated to require daytime oxygen therapy during the course of the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15185 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Participants with Symptomatic Mild, Moderate, or Severe Coronavirus Disease 2019 (COVID-19) | From Day 28 to Day 386
  Number of participants, testing serologically negative for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at baseline, with first occurrence of positive (+) polymerase chain reaction (PCR)-confirmed SARS-CoV-2 illness with symptomatic mild, moderate, or severe COVID-19 with onset from Day 28 through the length of the study.

SECONDARY OUTCOMES:
Participants with Symptomatic Moderate or Severe COVID-19 | From Day 28 to Day 386
  Number of participants, testing serologically negative for SARS-CoV-2 at baseline with first occurrence of (+) PCR-confirmed, SARS-CoV-2 illness with symptomatic moderate or severe COVID-19 with onset from Day 28 through the length of the study.
Participants with Symptomatic Severe COVID-19 | From Day 28 to Day 386
  Number of participants, testing serologically negative for SARS-CoV-2 at baseline with first occurrence of (+) PCR-confirmed, SARS-CoV-2 illness with symptomatic severe COVID-19 with onset from Day 28 through the length of the study.
Participants with Symptomatic Mild, Moderate, or Severe COVID-19 Regardless of Baseline Serostatus | From Day 28 to Day 386
  Number of participants, regardless of serostatus at baseline, with first occurrence of (+) PCR-confirmed, SARS-CoV-2 illness with symptomatic mild, moderate, or severe COVID-19 assessed from Day 28 through the length of the study.
Participants with Asymptomatic or Symptomatic COVID-19 | From Day 28 to Day 386
  Number of participants, regardless of serostatus at baseline, with first occurrence of (+) PCR-confirmed, or nucleocapsid protein serologically confirmed, SARS-CoV-2 illness with asymptomatic or symptomatic COVID-19 with onset from Day 28 through the length of the study.
Participants with COVID-19 requiring Hospitalization, Intensive Care Unit (ICU), or Mechanical Ventilation | From Day 28 to Day 386
  Number of participants, regardless of serostatus at baseline, with first occurrence of (+) PCR-confirmed, SARS-CoV-2 illness with COVID-19 with onset from Day 28 through the length of the study.
Participants with Symptomatic Mild COVID-19 | From Day 28 to Day 386
  Number of participants, regardless of serostatus at baseline, with first occurrence of (+) PCR-confirmed, SARS-CoV-2 illness with symptomatic mild COVID-19 (with no progression to moderate or severe COVID-19 during the course of the COVID-19 episode) with onset from Day 28 through the length of the study.
Serum IgG Antibody Levels at Multiple Time Points Expressed as Geometric Mean ELISA Units (GMEUs) | Day 0 to Day 35
  Serum IgG antibody levels specific for the SARS-CoV-2 rS protein antigen(s) as detected by enzyme-linked immunosorbent assay (ELISA) expressed as GMEUs at Day 0 and Day 35.
Participants with Serious Adverse Events (SAEs) | 386 days
  Number of participants with SAEs through the length of the study by Medical Dictionary for Regulatory Activities (MedDRA) classification and relationship to study vaccination.
Participants with Medically Attended Adverse Events (MAAEs) Related to Study Vaccination | 386 days
  Number of participants with MAAEs related to study vaccination through the length of the study by MedDRA classification.
Participants with Adverse Events of Special Interest (AESIs) | 386 days
  Number of participants with AESIs, which include potential immune-mediated medical conditions (PIMMCs) and AESIs relevant to COVID-19 such as possible vaccine-enhanced disease by MedDRA classification through the length of the study.
Participants with Solicited Local and Systemic Adverse Events (AEs) | 28 days
  Number of participants with solicited local and systemic AEs for 7 days after each study vaccination.
Participants with All MAAEs Through Day 35 | 35 days
  Number of participants with all MAAEs through Day 35 by MedDRA classification and relationship to study vaccination.
Participants with Unsolicited AEs Through Day 49 | 49 days
  Number of participants with unsolicited AEs through Day 49 by MedDRA classification and relationship to study vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.; Paul T Heath, MB BS FRACP FRCPCH, Principal Investigator — Vaccine Institute, St Georges, University of London
Locations (33):
- United Kingdom (33):
  - Belfast Health and Social Care Trust (BHSCT) (Site UK011), Belfast, Antrim
  - Synexus Midlands Clinical Research Centre (Site UK024), Edgbaston, Birmingham
  - The Royal Cornwall Hospitals NHS Trust (Site UK036), Truro, Cornwall
  - Royal Devon and Exeter Hospital (Site UK013), Exeter, Devon
  - "Maidstone Hospital - Central Research and Development Office Above Breast Care Centre - 1st Floor" (Site UK028), Maidstone, Kent
  - Queen Elizabeth University Hospital (Site UK008), Glasgow, Lanarkshire
  - Blackpool Teaching Hospitals (Site UK010), Blackpool, Lancashire
  - Salford Hospital (Site UK030), Oldham, Lancashire
  - Synexus Merseyside Clinical Research Centre (Site UK026), Waterloo, Liverpool
  - Royal Free (Site UK012), Hampstead, London
  - St. George's University Hospitals NHS Foundation Trust Clinical Research Facility (Site UK001), Tooting, London
  - North Wales Clinical Research Centre (NWCRC) (Site UK027), Wrexham, North Wales
  - Lakeside Healthcare, Lakeside Surgery (Site UK005), Corby, Northants
  - Warneford Hospital (Site UK016), Oxford, Oxfordshire
  - Aberdeen Royal Infirmary (Site UK007), Foresterhill, Aberdeen
  - Bradford Teaching Hospitals NHS Trust (Site UK018), Bradford
  - Synexus Wales Clinical Research Centre (Site UK025), Cardiff
  - Synexus Lancashire Clinical Research Centre (Site UK022), Chorley
  - Colchester Hospital (Site UK034), Colchester
  - AES - Glasgow (Site UK033), Glasgow
  - University Hartlepool Hospital (Site UK021), Hartlepool
  - Synexus Hexham Clinical Research Centre (Site UK023), Hexham
  - Royal Lancaster Infirmary (Site UK029), Lancaster
  - Research & Innovation Centre, St. James's University Hospital (Site UK019), Leeds
  - St. Thomas' Hospital (Site UK020), London
  - Chelsea & Westminster NHS Foundation Trust (Site UK006), London
  - AES - Synexus Manchester (Site UK032), Manchester
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norfolk and Norwich University Hospital (Site UK015), Norwich
  - Wansford and Kingscliffe Practice (Site UK035), Peterborough
  - AES - Synexus Thames Valley (Site UK031), Reading
  - University Hospital Southampton NHS Foundation Trust (UHS) (Site UK014), Southampton
  - Midlands Partnership NHS Foundation Trust Headquarters (Site UK017), Stafford
  - Stockport NHS Foundation Trust (Site UK009), Stockport

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toback S, Galiza E, Cosgrove C, Galloway J, Goodman AL, Swift PA, Rajaram S, Graves-Jones A, Edelman J, Burns F, Minassian AM, Cho I, Kumar L, Plested JS, Rivers EJ, Robertson A, Dubovsky F, Glenn G, Heath PT; 2019nCoV-302 Study Group. Safety, immunogenicity, and efficacy of a COVID-19 vaccine (NVX-CoV2373) co-administered with seasonal influenza vaccines: an exploratory substudy of a randomised, observer-blinded, placebo-controlled, phase 3 trial. Lancet Respir Med. 2022 Feb;10(2):167-179. doi: 10.1016/S2213-2600(21)00409-4. Epub 2021 Nov 17. PMID 34800364
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: CDC (Centers for Disease Control and Prevention): Coronavirus (COVID-19) website — http://www.CDC.gov/coronavirus/2019-nCoV/index.html
- See also: WHO COVID-19 treatment guidelines — http://www.who.int/emergencies/diseases/novel-coronavirus-2019/
- See also: NHS Health Research Authority: COVID-19 Research — https://www.hra.nhs.uk/covid-19-research/